CLINICAL TRIAL: NCT04773158
Title: Systematic Pediatric Assessment of Rome Criteria
Brief Title: Systematic Pediatric Assessment of Rome Criteria (SPARC)
Acronym: SPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William E. Bennett, Jr., Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1811325201; R01DK118433 (NIH)
Record Dates: First submitted 2020-05-11; First posted 2021-02-26 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: Computerized Decision Support
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Will perform cluster randomization by clinic. The unit of randomization will be the clinic site, but the unit of analysis will be the individual patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention clinic sites will be provided access to both the Functional gastrointestinal disorders (FGIDs) Screening Module and the Treatment Module
  Interventions: Behavioral: Clinical Decision Support
- Control Arm (No Intervention): The control clinics will have the Functional gastrointestinal disorders (FGIDs) Screening Module. However, control clinics will not have access to the FGIDs Treatment Module. These clinic sites will be given access to the pre-screener form section of the module, so that providers are made aware of a positive screen for a FGID.

INTERVENTIONS:
Behavioral: Clinical Decision Support — The intervention clinic sites will be provided access to a Clinical Decision Support System (CDSS) that incorporates the Rome IV criteria for evidence-based care recommendations for functional gastrointestinal disorders (FGIDs)
  Arms: Intervention Arm

SUMMARY:
While gastroenterologists care for many of the pediatric patients with Functional gastrointestinal disorders (FGIDs), the majority of the burden continues to be borne by general pediatricians, especially with respect to initial diagnosis. Unfortunately, FGIDs are often diagnosed incorrectly by primary care providers, and patients often wait months to years before a correct diagnosis is made, and effective treatment is begun. Furthermore, primary care providers are often unaware of recent guideline changes or the evidence base for children with FGIDs, leading to overuse of testing, inappropriate or ineffective treatment, and increased costs. Given this information, it is essential that we develop interventions that target pediatric primary care providers to improve their care for children with FGIDs. The investigators propose that using a Clinical Decision Support System (CDSS) that incorporates the Rome IV criteria for diagnosis and evidence-based care for FGIDs will improve the (1) accuracy of diagnosis and (2)_ effectiveness of clinical care. A CDSS has advantages with respect to guideline adherence and automated diagnosis, because it can provide focused, real-time, patient-specific data to the clinician. The investigators hypothesize that automation of screening, diagnosis, and management of FGIDs using the Rome IV criteria will result in improved resolution of FGIDs (primary outcome), as well as decreased utilization of medical services (secondary outcomes). This hypothesis will be tested utilizing a randomized controlled trial. The intervention clinic sites will be provided access to both the FGIDs Screening Module and the Treatment Module. The control clinics will have the FGIDs Screening Module. However, control clinics will not have access to the FGIDs Treatment Module. These clinic sites will be given access to the pre-screener form section of the module, so that providers are made aware of a positive screen.

DETAILED DESCRIPTION:
Functional gastrointestinal disorders (FGIDs) are extremely common in children and adolescents, and represent a wide range of disorders that are related to the gastrointestinal tract, but have no clear structural, anatomic, or histopathologic cause. FGIDs represent an enormous burden on patients and families, and patients with these functional disorders have much higher health care utilization and related costs. As there are no biochemical markers or structural abnormalities that can be used to diagnose these disorders in children objectively, FGIDs are diagnosed according to the symptom-based Rome criteria. While gastroenterologists care for many of the pediatric patients with FGIDs, the majority of the burden continues to be borne by general pediatricians, especially with respect to initial diagnosis. Unfortunately, FGIDs are often diagnosed incorrectly by primary care providers, and patients often wait months to years before a correct diagnosis is made, and effective treatment is begun. Furthermore, primary care providers are often unaware of recent guideline changes or the evidence base for children with FGIDs, leading to overuse of testing, inappropriate or ineffective treatment, and increased costs. Given this information, it is essential to develop interventions that target pediatric primary care providers to improve their care for children with FGIDs. This study proposes that using a Clinical Decision Support System (CDSS) that incorporates the Rome IV criteria for diagnosis and evidence-based care for FGIDs will improve the (1) accuracy of diagnosis and (2)_ effectiveness of clinical care. A CDSS has advantages with respect to guideline adherence and automated diagnosis, because it can provide focused, real-time, patient-specific data to the clinician. Studies of barriers to guideline implementation have shown multiple factors at work: unfamiliarity with a guideline, lack of self-efficacy, or difficulty implementing the guideline components within the current workflow of a practice. CDSS can overcome many of these barriers because they are integrated with systems that routinely store and retrieve patient information and can improve workflow by providing clinicians with patient-specific advice at the time of the patient visit. The study investigators hypothesize that automation of screening, diagnosis, and management of FGIDs using the Rome IV criteria will result in improved resolution of FGIDs (primary outcome), as well as decreased utilization of medical services (secondary outcomes). This hypothesis will be tested utilizing a randomized controlled trial. The intervention clinic sites will be provided access to both the FGIDs Screening Module and the Treatment Module. The control clinics will have the FGIDs Screening Module. However, control clinics will not have access to the FGIDs Treatment Module. These clinic sites will be given access to the pre-screener form section of the module, so that providers are made aware of a positive screen for a FGID. The investigators have chosen not to have an arm without provider notification due to concern that identification of symptoms without notifying the patient's provider represented an ethical concern. If anything, this will bias towards a null result. Since FGIDs have both a high rate of relapse, and a high rate of spontaneous resolution, it is necessary to assess the pattern of symptoms across multiple time points. As such, we plan to gather various data from parents/patients at 1, 3, 6 and 12-months via phone interview. Additionally, the study will assess parental satisfaction with the screening and treatment of their child's particular FGID at the 3-month phone interview. For assessment of health care utilization, the study will look at the following variables in the 12 months after initial Rome IV screening positive: a) outpatient sick visits for any complaint; b) outpatient sick visits with an associated GI billing code; c) visits to statewide providers, including inpatient hospital stays, outpatient clinic visits, and emergency room visits; d) GI-related testing and procedures; e) use of any medications prescribed to treat Rome IV diagnoses. These data will be obtained from multiple sources including the EMR, and Indiana Network for Patient Care (INPC).

ELIGIBILITY:
Inclusion Criteria:

* Any patient between the ages of 0 through 17 presenting to a pediatric primary care clinic in the Eskenazi health system and the Primary Care Physician who sees them

Exclusion Criteria:

* None

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2025-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Bennett, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Clinical Sites
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 21; 4 Clinical Sites | 12; 4 Clinical Sites
Completed | 17; 4 Clinical Sites | 10; 4 Clinical Sites
Not Completed | 4; 0 Clinical Sites | 2; 0 Clinical Sites

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 21 | 12 | 33
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 7.9 [4.05 to 12.8] | 7.2 [2.35 to 9.3] | 7.9 [3.2 to 12.15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 12 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 18 | 7 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 13 | 4 | 17
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 21 | 12 | 33

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Symptoms From Initial Rome IV Diagnosis at 3 Months Using an Age-appropriate Rome IV Questionnaire. Number of Participants Who no Longer Meet Rome IV Criteria.
Description: This measure will be determined for the Rome IV diagnoses of: Aerophagia, Rumination, Functional Constipation, Cyclic Vomiting Syndrome (CVS), Functional Diarrhea, Non Retentive Fecal Incontinence, Functional Vomiting, Functional Nausea, Functional Dyspepsia- Postprandial Distress Subtype, Functional Dyspepsia- Epigastric Pain Syndrome Subtype, Irritable Bowel Syndrome (IBS), Abdominal Pain otherwise Not Specified, and Abdominal Migraine. The presence or absence of meeting criteria for the Rome IV diagnoses will be coded as a binary variable (true/false) to represent resolution of symptoms.
Time Frame: 3 months from initial diagnosis
Population: Results reflect the number of participants who no longer met Rome IV Criteria coded as a binary variable "False". Of the 21 enrolled, 20 patients in the intervention group and 11 patients in the control group had a diagnosis within the Rome IV diagnoses listed. For the intervention arm, 18 of the 20 participants completed the 3 month questionnaire. For the control arm, 5 of 11 participants completed the 3 month questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 18 | 5
Participants | 17 | 3

2. Primary Outcome: Change in Parental Concern for the Rome IV Diagnoses of Infant Regurgitation, Infant Dyschezia, and/or Infant Colic From Initial Rome IV Diagnosis at 3 Months Using Likert Scale Questionnaire. Number of Participants With Ongoing Concern.
Description: This change will be measured by a single likert scale question asked in the FGID Screening module (Baseline) and again at the 3 month follow up phone survey. , The parent is able to indicate their degree of concern about the symptomology associated with the Rome IV diagnosis. The presence or absence of ongoing concern will then be coded as a binary variable (true/false).
  Likert scale: Not at all concerned, Slightly concerned, Somewhat concerned, Moderately concerned, Extremely concerned
Time Frame: Baseline and 3 months from initial diagnosis
Population: Results reflect the number of participants with the presence of ongoing concern, coded as a binary variable true. Of 21 enrolled, 1 in the intervention group and 1 in the control group had a diagnosis within the Rome IV diagnoses listed. For each arm, 1 of 1 completed the 3 month questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

3. Secondary Outcome: Resolution of Symptoms From Initial Rome IV Diagnosis at 1, 6 and 12 Months Using an Age-appropriate Rome IV Questionnaire.
Description: as for outcome 1
Time Frame: 1, 6 and 12 months from initial diagnosis
Reporting Status: Not Posted

4. Secondary Outcome: Change in Parental Concern (for the Rome IV Diagnoses of Infant Regurgitation, Infant Dyschezia, and/or Infant Colic From Initial Rome IV Diagnosis at 1 an 6 Months Using Likert Scale Questionnaire
Description: as for outcome 2
Time Frame: 1 and 6 months from initial diagnosis
Reporting Status: Not Posted, anticipated posting 2025

5. Secondary Outcome: Parent Satisfaction With Screening Measured at 3 Months Using a Likert Scale Questionnaire [Very Dissatisfied , Dissatisfied, Unsure, Satisfied, Very Satisfied]
Description: This was measured by two likert scale questions asked in the 3 month follow up phone call.
Time Frame: 3 months from initial diagnosis
Population: For intervention arm, 14 of 21 participants enrolled completed this questionnaire. For the control arm, 8 of 12 participants enrolled completed this questionnaire.
Measure: Number; unit: participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 14 | 8
participants
  Very dissatisfied | 0 | 0
  Dissatisfied | 1 | 0
  Unsure | 3 | 1
  Satisfied | 5 | 5
  Very satisfied | 5 | 2

6. Secondary Outcome: Parent Satisfaction With Treatment Measured at 3 Months Will be Measured Using a Likert Scale Questionnaire [Very Dissatisfied , Dissatisfied, Unsure, Satisfied, Very Satisfied]
Description: This will be measured by two likert scale questions asked in the 3 month follow up phone call. Satisfaction with screening and treatment of FGID will be assessed.
Time Frame: 3 months from initial diagnosis
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 14 | 8
participants
  Very dissatisfied | 0 | 0
  Dissatisfied | 0 | 1
  Unsure | 5 | 4
  Satisfied | 4 | 2
  Very satisfied | 5 | 1

7. Secondary Outcome: Rate of Health Care Utilization Will be Assessed 12 Months After Initial Rome IV Screening Positive. Variables Will be Coded as Binary Variables (True/False)
Description: The following variables will be assessed: Outpatient sick visits for any complaint, Outpatient sick visits with an associated GI billing code; Visits to statewide providers, including inpatient hospital stays, outpatient clinic visits, and emergency room visits; The occurrence of any GI-related testing and procedures - specifically radiologic, laboratory testing, endoscopy, and surgical procedures related to GI diagnoses; The use of any medications prescribed to treat Rome IV diagnoses - specifically acid- suppressants, antispasmodics, antidepressants, stool softeners and laxatives, and pro-motility agents
Time Frame: 12 months from initial diagnosis
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Description: Nov 22, 2021-Feb 6, 2025 Adverse event data was monitored from enrollment of first patient to last data collection point on last patient
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/12
Other Adverse Events (participants affected / at risk) | 0/21 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT04773158/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04773158/SAP_001.pdf
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT04773158/ICF_002.pdf